CLINICAL TRIAL: NCT04912323
Title: The R3 Vascular Drug-Eluting Bioresorbable Scaffold in Below the Knee Vessels Trial (RESOLV I)
Brief Title: Study of the R3 Vascular Drug-Eluting Bioresorbable Scaffold in Treating Below the Knee Arterial Disease
Acronym: RESOLV I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: R3 Vascular Inc. (Industry)
Collaborators: Massachusetts General Physicians Organization / Vascore (Unknown); Cardiovascular Research Foundation, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-1501
Record Dates: First submitted 2021-05-18; First posted 2021-06-03 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Peripheral Arterial Disease; Atherosclerotic Lesion; Lower Extremity Ischemia; Lower Extremity Claudication
Keywords: Claudication; Leg Pain; Lower Extremities; Lower Limb; Blocked Leg Artery; Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Intervention Model Description: All subjects will receive the investigational device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- MAGNITUDE® Scaffold (Experimental): Subject with up to three study lesions treated by implanting a maximum of 3 R3 Vascular MAGNITUDE® Bioresorbable Drug-Eluting Scaffolds
  Interventions: Device: Percutaneous Implantation of the MAGNITUDE® Bioresorbable Arterial Scaffold

INTERVENTIONS:
Device: Percutaneous Implantation of the MAGNITUDE® Bioresorbable Arterial Scaffold — Placement of one or more MAGNITUDE® bioresorbable scaffolds using a percutaneous technique at one or more arterial stenoses.

SUMMARY:
This first-in-human clinical feasibility study will evaluate the safety and performance of the R3 Vascular MAGNITUDE® Bioresorbable Drug-Eluting Scaffold and Delivery System in patients undergoing treatment for peripheral arterial disease severe enough to have significantly reduced the blood supply to their leg. The severe reduction in blood flow causes lifestyle limiting leg pain for these patients, and may lead to amputation of the affected limb due to the loss of tissue in the leg or foot from ulcers or gangrene. The investigational device being studied in this trial is intended to restore blood flow to the affected limb, providing symptomatic relief to the patient and reducing the risk of limb amputation. The scaffold is a type of vascular stent placed within the diseased artery below the knee to improve blood flow. Unlike commercially available metallic stents which are permanently placed within the artery, the MAGNITUDE® Bioresorbable scaffold is made of a polymer material that will completely dissolve away over time, providing the support necessary to the artery while it is healing after the treatment procedure and then slowly disappearing from the artery once that support is no longer needed. The investigational scaffold has been successfully used to treat vascular blockages in the coronary arteries of the heart, but the RESOLV I study will be the first time this device has been used to improve blood flow in the arteries of the lower leg. Patients enrolled in this study may have up to three vascular blockages in their lower leg arteries treated with the MAGNITUDE® Bioresorbable scaffold, and then will be assessed over the course of the following five years to evaluate whether the investigational treatment was successful in safely alleviating their leg pain and other symptoms.

DETAILED DESCRIPTION:
The prevalence of peripheral artery disease (PAD) is estimated to be over 200 million. Critical limb ischemia (CLI) is considered the most advanced stage of PAD, occurring in about 10% of PAD patients. CLI patients typically present with ischemic rest pain, nonhealing ulcerations, infection, and/or gangrene. It is associated with a high risk of major amputation (lower limb amputations in 10% - 40% of patients at 6 months), cardiovascular events, and death (mortality rate of 20% within 6 months after the diagnosis and 50% at 5 years). A large percentage of CLI patients have occlusive disease in the infrapopliteal artery, especially in diabetics where PAD is 3 - 4 times more common. CLI related to diabetes is often more extensive, with multiple long segmental occlusions resulting in a 5 - 30-fold increase in the rate of amputations. Surgical and catheter-based revascularization procedures are typically performed to restore distal perfusion and prevent amputation in symptomatic patients.

Surgical bypass has been shown to be an effective treatment when anatomic and patient risk factors permit this approach. However, patients with CLI are often poor surgical candidates because of the absence of suitable graft vessels or the presence of significant medical comorbidities. During the past decade, therapies such as percutaneous transluminal angioplasty (PTA) and percutaneous treatment with balloons or the off-label use of coronary stents that deliver antiproliferative drugs directly to the vessel wall to inhibit neointimal hyperplasia have been on the rise and have decreased the rates of open bypass surgery.

Percutaneous transluminal angioplasty has become the first line revascularization therapy for patients with symptomatic peripheral artery disease. Published literature indicates that while uncoated balloon angioplasty has a high rate of technical success in obtaining a patent lumen, restenosis requiring repeat revascularization or amputation is common. For femoropopliteal (above the knee) disease, percutaneous treatment with a balloon that delivers an antiproliferative agent (usually paclitaxel) directly to the vessel wall inhibits neointimal hyperplasia and significantly reduces the rate of target lesion revascularization and restenosis, while maintaining a safety profile comparable to that of uncoated balloons. On the other hand, drug-coated balloon (DCB) therapy in the infrapopliteal (below the knee) arteries has not shown similarly convincing evidence of superiority over PTA, and in general, the use of DCB below the knee remains controversial.

Metallic drug-eluting stents have been shown to effective in reducing both abrupt vessel closure and restenosis rates in the management of peripheral vascular disease. However, metallic implants also negatively impact the vessel wall by permanently preventing vasomotion, autoregulation, and adaptive remodeling. In addition, there is a risk of late vessel failure due to incomplete endothelialization of the implant, stent fracture, or malapposition. Metallic implants may also cause artifacts with noninvasive imaging and complicate future revascularization procedures. Bioresorbable scaffolds provide similar mechanical properties to metallic stents during the blood vessel remodeling phase following angioplasty, while also delivering an antiproliferative drug to the site of vascular injury to minimize neointimal hyperplasia. However, once these tasks are complete, the scaffold begins a reabsorption process and eventually disappears entirely from the vessel, leaving the native artery free of any implant. For these reasons, bioresorbable scaffolds may offer a new standard for restorative therapy in the peripheral vasculature.

This first-in-human clinical feasibility study of the R3 Vascular MAGNITUDE® scaffold will evaluate the safety and performance of a bioresorbable scaffold with a thin strut design (98 µm wall thickness) and a coating of the antiproliferative drug Sirolimus for treating patients with lifestyle limiting claudication or chronic limb threatening ischemia. The objective is to perform an initial evaluation of the investigational device in a patient population undergoing percutaneous transluminal intervention with stenting for the treatment of infrapopliteal artery lesions.

The thin strut design of the MAGNITUDE® scaffold offers improved deliverability and the potential for higher vessel patency rates compared to other thicker strut bioresorbable scaffolds currently under investigation for this particular indication. In addition, compared with metallic stents, the R3 Vascular bioresorbable scaffold provides sustained support to the vessel wall following revascularization while vascular healing occurs, after which the scaffold predictably degrades leaving no permanent implant behind. The MAGNITUDE® scaffold has been shown to be biocompatible, maintain mechanical integrity over time, and provide controlled drug release through extensive validations in pre-clinical testing and clinical studies enrolling approximately 200 patients being treated for coronary artery disease.

The RESOLV I clinical investigation is a prospective, single-arm, multi-center first-in-human feasibility study of the R3 Vascular MAGNITUDE® Bioresorbable Drug-Eluting Scaffold and Delivery System for treating vascular disease in the infrapopliteal arteries. It will enroll a maximum of 30 patients from up to 9 investigational centers in Italy, Austria, and Canada. Eligible patients who are at least 18 years of age with lifestyle limiting claudication or chronic limb threatening ischemia (Rutherford-Becker categories 3 - 5) that elect to undergo revascularization with stenting of up to three different de novo or restenotic infrapopliteal artery lesions will be treated with the investigational device and followed for five years post-implantation.

Safety of the investigational scaffold will be assessed at 6 months as the composite rate of Major Adverse Limb Events (above ankle amputation in the index limb or major re-intervention) and peri-operative (30-day) mortality. Performance of the device will be evaluated as the primary patency rate of the treated vessels at 6 months, assessed by angiography. Multiple other angiographic, duplex ultrasound, and clinical assessments will be performed during the 5-year follow-up period.

It is expected that the subjects enrolled in this study will experience the same benefits as patients treated with the currently available coronary (used off label in the peripheral arteries) drug-eluting metallic stents. Treatment with the investigational scaffold may provide physicians with a promising alternative to permanent stenting, which has been shown to interfere with future treatments such as PTA or surgery. Additionally, since the investigational scaffold is designed to provide mechanical support to the target lesion for the required healing period post-treatment and disappear once healing is complete, this may allow for positive remodeling of the artery and reduce the risk of late complications (i.e., endothelial cell proliferation, restenosis, thrombosis, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years and ≤ 90 years of age.
* Subject agrees not to participate in any other investigational device or drug study for a period of at least six months following the index procedure. Questionnaire-based studies, or other studies that are non-invasive and do not require investigational devices or medications are allowed.
* Subject (or their legally authorized representative) provides written informed consent prior to any study-related procedure, using the form approved by the local Ethics Committee.
* Subject has lifestyle limiting claudication or chronic limb threatening ischemia (Rutherford-Becker categories 3 - 5).
* Subject agrees to complete all protocol required follow-up visits, including angiograms.
* Subject has suitable common femoral (contralateral or antegrade ipsilateral) vascular access. (Note: Radial or pedal access not allowed.)
* Subject has up to three de novo or restenotic native infrapopliteal lesions with > 70% stenosis by angiography.
* Lesion(s) must be located in the proximal 2/3 of native infrapopliteal vessels and at least 10 cm above the tibio-talar joint.
* Reference vessel(s) diameter of 2.5 - 3.5 mm by IVUS.
* A maximum of three 18 mm scaffolds, or one 38 mm scaffold, or one 18 mm length scaffold with one 38 mm length scaffold can be implanted per patient.
* Scaffold(s) must cover at least 2 mm from the pre-dilatation borders, resulting in a maximum allowed lesion length of:

  1. 14 mm for a single 18 mm length scaffold
  2. 31 mm for two overlapping 18 mm length scaffolds (using the marker overlap technique)
  3. 47 mm for three overlapping 18 mm length scaffolds (using the marker overlap technique)
  4. 34 mm for a single 38 mm length scaffold
  5. 51 mm for a single 38 mm length scaffold with a single overlapping 18 mm length scaffold (using the marker overlap technique)
* Tandem non-contiguous lesions, if present, having plaque-free zones between the lesions of ≥ 2 cm can be treated with any combination of up to three scaffolds (1-1-1, 1-2, or 2-1).
* Lesion (most distal lesion if more than one is being treated) must be successfully crossed in antegrade fashion with a guidewire. (Note: The most distal lesion should be treated before treating more proximal lesions.)
* Target lesion(s) preparation prior to scaffold placement with non-compliant balloon (1:1 balloon:artery ratio) must achieve < 50% residual diameter stenosis by angiography. (Note: The use of specialty balloons such as cutting, scoring, serration, or the Chocolate PTA balloon in 1:1 balloon:artery ratio is allowed if required lesion preparation not achieved with the initial non-compliant balloon. Atherectomy is not allowed.)
* Inflow above-the-knee lesions (> 50% diameter stenosis by angiography), if present, must be treated successfully using the standard of care per site prior to target lesion(s). (Note: Inflow lesions may be treated during the index procedure.)
* Non-target below-the-knee lesions in other non-target vessels, if present, may be treated at the discretion of the investigator per standard of care, but must be treated successfully prior to the target lesion(s).
* At least one fully patent below-the-ankle artery (i.e., dorsalis pedis; common, lateral, or medial plantar arteries) without hemodynamically significant lesions (≥ 50% diameter stenosis by angiography) must be present in the target limb.

Exclusion Criteria:

* Pregnant or nursing subjects and those who plan pregnancy within 6 months following index procedure. (Note: Subjects of child-bearing potential must have a negative pregnancy test ≤ 28 days prior to the index procedure and agree to use contraception for 6 months.)
* Presence of other significant comorbid conditions, or other medical, social, or psychological conditions (such as history of substance {alcohol, cocaine, heroin, etc.} abuse), that in the investigator's opinion may limit the subject's ability to participate or comply with study instructions and follow-up (includes subjects with symptomatic COVID-19 infection in the past 2 months or asymptomatic COVID-19 positive test in the past 1 month).
* Incapacitated individuals, defined as persons who are mentally ill, mentally handicapped, or individuals without legal authority to control their activities.
* Life expectancy of < 1 year.
* Subject is non-ambulatory.
* Subject has prior major amputation (either limb).
* Subject has chronic renal insufficiency stage 4 or above or requires dialysis.
* Subject has known hypersensitivity or contraindication to device materials and their degradants (sirolimus, poly (L-lactide), poly (D, L-lactide), lactic acid, or platinum-iridium) or to study medications (including antiplatelet medications) or to contrast media and who cannot be adequately premedicated.
* Subject with planned surgery or procedure necessitating discontinuation of antiplatelet medications within 6 months after the index procedure.
* Subject has active systemic infection.
* Subject has a prior stroke or MI within 3 months of the index procedure.
* Subject has presence of osteomyelitis or any gangrene above the metatarsal-phalangeal joints, extensive tissue loss with exposed tendons or requiring complex or recurrent surgeries, full thickness heel ulcer, or pure neuropathic ulcers.
* Subject is receiving immunosuppression therapy and/or has known immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus, rheumatoid arthritis, severe asthma requiring immunosuppressive medication, etc.).
* Subject has active malignancy (receiving or scheduled to receive anticancer therapy for malignancy within 1 year prior to or after the index procedure), active blood dyscrasia or coagulation disorder (platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a WBC < 3,000 cells/mm3, or hemoglobin < 8.0 g/dl).
* Subject with uncontrolled diabetes with HbA1c > 10%.
* Subject with Body Mass Index (BMI) < 18.
* Revascularization procedure within the target vessel in the previous 3 months.
* Planned surgical or endovascular procedures within 30 days. (Note: A planned minor amputation is allowed.)
* The target vessel(s) have any other distal hemodynamically significant lesions (≥ 50% diameter stenosis by angiography).
* Lesions in which successful predilation cannot be achieved.
* Target lesion location requires bifurcation treatment method that requires scaffolding of both branches (provisional treatment, without the need of scaffolding use in a side branch is acceptable).
* Presence of aneurysm or acute thrombus in the aorta or lower extremity arteries.
* Prior below-the-knee bypass in the target limb.
* Previously stented lesion(s) or the presence of stents in the target vessel.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
(Safety) Freedom from MALE and POD | MALE is assessed at 180 days and POD is assessed at 30 days (post implantation procedure)
  Composite endpoint of freedom from Major Adverse Limb Event ("MALE", which includes above ankle amputation in the index limb or major re-intervention) and Peri-Operative Death ("POD")
(Performance) Primary Patency of the Target Lesion(s) | Assessed at 180 days (post implantation procedure)
  Freedom from hemodynamically significant stenosis by angiography (≥ 50% diameter stenosis), or duplex ultrasound (absence of flow per core lab) when angiography is not available, without additional target lesion revascularization

SECONDARY OUTCOMES:
Technical Success | Assessed from start of treatment procedure to end of treatment procedure
  Defined as delivery and deployment of the scaffold to the target lesion resulting in a final angiographic in-lesion percent diameter stenosis ≤ 30%
Procedural Success | Assessed from start of treatment procedure to hospital discharge after treatment procedure, approximately same day or day after treatment procedure
  Defined as Technical Success without procedural Major Adverse Event (which includes thrombosis, distal embolization, or vessel rupture)
Angiographic Acute Gain | Assessed at 180 days (post implantation procedure)
  Defined as the difference between the post- and pre-procedural minimal lumen diameter within the scaffold and within the scaffolded vessel segment as assessed by angiography
Angiographic Late Lumen Loss | Assessed at 180 days (post implantation procedure)
  Defined as the difference between the post-procedural and follow-up minimal lumen diameter within the scaffold and within the scaffolded vessel segment as assessed by angiography
Angiographic Binary Restenosis | Assessed at 180 days (post implantation procedure)
  Defined as a > 50% diameter stenosis within the scaffold and within the scaffolded vessel segment at follow-up as assessed by angiography
Duplex Ultrasound Detection of Arterial Flow | Assessed at 1, 6, and 12 months (post implantation procedure)
  Determination of the presence or absence of blood flow within the target lesion(s) and vessel(s)
All-Cause Death | Assessed at 1, 3, 6, 12, 24, 36, 48 and 60 months (post implantation procedure)
  Defined as patient mortality due to any cause
Clinically Driven Target Lesion Revascularization | Assessed at 1, 3, 6, 12, 24, 36, 48 and 60 months (post implantation procedure)
  Defined as revascularization for a target lesion if the target lesion diameter stenosis is > 70% by angiography, or > 50% and the subject has ischemia that cannot be explained by another lesion, or ≤ 50% if severe ischemic signs are attributable to the target lesion.
Freedom from Composite of Target Lesion Occlusion, Clinically Driven Target Lesion Revascularization, and Major Amputation | Assessed at 1, 3, 6, 12, 24, 36, 48 and 60 months (post implantation procedure)
  Subject has not experienced occlusion of the target lesion necessitating revascularization due to ischemic symptoms or amputation of the target limb.
Change in Rutherford-Becker Classification from Enrollment | Assessed at 1, 3, 6, 12, 24, 36, 48 and 60 months (post implantation procedure)
  Change between the pre-treatment and follow-up assessments of the symptomatic classification of the subject's chronic limb ischemia
Change in Ankle-Brachial Index (ABI) from Enrollment | Assessed at 1, 3, 6, and 12 months (post implantation procedure)
  Change between the pre-treatment and follow-up assessments of the comparison of the blood pressure measured at the ankle with the blood pressure measured at the arm to gauge the degree of arterial narrowing in the leg
Change in Toe-Brachial Index (TBI) from Enrollment | Assessed at 1, 3, 6, and 12 months (post implantation procedure)
  Change between the pre-treatment and follow-up assessments of the comparison of the blood pressure measured at the toes with the blood pressure measured at the arm to gauge the degree of arterial narrowing in the leg

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Granada, MD, Principal Investigator — Cardiovascular Research Foundation (CRF)
Locations (7):
- Medical University Graz, Graz, Austria
- Canada (3):
  - CRCHUM Université Montreal, Montreal
  - Hopital Saint-Francois d'Assise, Québec
  - Toronto General Hospital, Toronto
- Italy (3):
  - San Donato Hospital, Arezzo
  - Maria Cecilia Hospital, Cotignola
  - IRCCS Multimedica, Milan

IPD SHARING:
Plan to Share IPD: No